CLINICAL TRIAL: NCT05043922
Title: A Phase II, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of CYH33, a Selective PI3Kα Inhibitor in Patients With Recurrent/Persistent Ovary, Fallopian Tube or Primary Peritoneal Clear Cell Carcinoma
Brief Title: A Study to Evaluate the Efficacy and Safety of CYH33 in Patients With Recurrent/Persistent Ovary Clear Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYH33-G201
Record Dates: First submitted 2021-08-30; First posted 2021-09-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Recurrent Cancer
Keywords: Phase 2 study; Pharmacokinetics
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — CYH33

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CYH33 (Experimental): 40mg daily
  Interventions: Drug: CYH33

INTERVENTIONS:
Drug: CYH33 — a Selective PI3Kα Inhibitor

SUMMARY:
The purpose of this study is to determine the treatment efficacy of CYH33 monotherapy in patients with recurrent or persistent ovarian, fallopian tube or primary peritoneal clear cell carcinoma harboring PIK3CA hotspot mutation, who received prior systemic anti-tumor treatment.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether treatment with single agent CYH33 significantly improves ORR compared to historical efficacy data in patients with recurrent/persistent ovarian clear cell carcinoma (OCCC) harboring PIK3CA hotspot mutations who received prior systemic anti-tumor treatment.

ELIGIBILITY:
Main Inclusion Criteria:

1. Female patients ≥ 18 years of age
2. Provide informed consent voluntarily.
3. Patients must have histologically or cytologically confirmed recurrent or persistent ovarian, fallopian tube, or peritoneum clear cell carcinoma.
4. Patients with recurrent/persistent ovary, fallopian tube or primary peritoneal clear cell carcinoma, who have identified PIK3CA status.
5. Patients must have failed standard chemotherapy.
6. ECOG-PS ≤ 1.
7. Patient must have adequate organ and bone marrow function measured within 28 days of screening.

Main Exclusion Criteria:

Patients are ineligible for this study if they meet any of the following criteria:

1. Patient has received any anticancer therapy
2. Patients who had prior treatment with any PI3K, mTOR or AKT inhibitor.
3. Radical radiation therapy within 4 weeks prior to the first dose of the investigational product or received local palliative radiation therapy for bone metastases within 2 weeks.
4. Any toxicities from prior treatment that have not recovered to baseline.
5. Patients who have been treated with any hematopoietic colony-stimulating growth factors ≤ 2 weeks prior to starting study drug.
6. Patients who have symptomatic CNS metastasis.
7. Major surgery or had significant traumatic injury within 28 days prior to the first dose of the investigational product or has not recovered from major side effects.
8. Known HIV infection with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunity infection within the past 12 months; active hepatitis B and hepatitis C.
9. History of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis.
10. Patients with clinically significant cardiovascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Tumor ORR in patients with PIK3CA hotspot mutations. | through study completion, an average of 1 year
  Tumor ORR per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 in patients with PIK3CA hotspot mutations.

SECONDARY OUTCOMES:
PFS | through study completion, an average of 1 year
  PFS by BIRC using RECIST v1.1
OS | through study completion, an average of 2 year
  OS in each of the PIK3CA mutation status cohort
genetic and protein biomarker alterations | through study completion, an average of 1 year
  genetic and protein biomarker alterations that can impact PI3K signaling pathway

OTHER OUTCOMES:
Safety and tolerability | through study completion, an average of 1 year
  type, incidence, duration, severity and seriousness of adverse events (AEs)
DLT (Dose Limiting Toxicity) in Japanese patients | 4 weeks
  Number and proportion of patients who experienced DLT during the first 28-day of treatment in Japanese patients in safety run-in study.
Peak Plasma Concentration (Cmax) | 4weeks
  Pharmacokinetics parameters
Area under the plasma concentration versus time curve (AUC) | 4weeks
  Pharmacokinetics parameters

CONTACTS AND LOCATIONS:
Locations (36):
- China (25):
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing
  - Chinese PLA General Hospital, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Southwest Hospital of AMU, Chongqing
  - Sun Yat-sen University Cancer Center, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangdong
  - The First Affiliated Hospital of Hainan Medical College, Haikou
  - The Third People's Hospital of Hainan Province, Hainan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Hubei Cancer Hospital, Hubei
  - Hunan Cancer Hospital, Hunan
  - Qilu Hospital of Shandong University, Jinan
  - Jiangsu Province Hospital, Nanjing
  - The People's Hospital Of Guangxi Zhuang Autonomous Region, Nanning
  - Qingdao Central Hospital, Qingdao
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai
  - Shanghai First Maternity and Infant Hospital, Shanghai
  - Xiaohua wu, Shanghai
  - West China Second University Hospital, Sichuan University, Sichuan
  - Tianjin Medical University General Hospital, Tianjin
  - Zhongnan Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Sir Run Run Shaw Hospital， School of Medicine, Zhejiang University, Zhejiang
- Japan (11):
  - Kurume University Hospital, Kurume, Fukuoka
  - Osaka University Hospital, Suita, Osaka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Jikei University Hospital, Minato-Ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Shikoku Cancer Center, Matsuyama
  - Nagoya University Hospital, Nagoya
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai

IPD SHARING:
Plan to Share IPD: No